CLINICAL TRIAL: NCT03667443
Title: The Effects of Myo-inositol Plus Alpha-lactalbumin in Ovulation Induction of PCOS Myo-inositol-resistant Patients
Brief Title: Myo-inositol Plus Alpha-lactalbumin in PCOS Myo-inositol-resistant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MILA
Record Dates: First submitted 2018-08-01; First posted 2018-09-12 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2023-01

CONDITIONS: PCOS; Myo-inositol-resistance
Keywords: myo-inositol; alpha-lactalbumin; polycystic ovary syndrome; anovulation; infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Infertility | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myo-inositol plus folic (Active Comparator)
  Interventions: Dietary Supplement: Myo-inositol + folic a.
- Myo-inositol + folic a. + α-lactalbumin (Active Comparator)
  Interventions: Dietary Supplement: Myo-inositol + folic a. + α-lactalbumin

INTERVENTIONS:
Dietary Supplement: Myo-inositol + folic a. + α-lactalbumin — 3 months of treatment
  Other Names: Inofolic HP
  Arms: Myo-inositol + folic a. + α-lactalbumin
Dietary Supplement: Myo-inositol + folic a. — 3 months of treatment
  Other Names: Inofolic
  Arms: Myo-inositol plus folic

SUMMARY:
The investigator's aim is to evaluate if the combination of myo-inositol and alpha-lactalbumin can overcome the resistance to myo-inositol in PCOS patients

DETAILED DESCRIPTION:
In this study, the investigators expect about 30% of the PCOS patients enrolled to be resistant to Myo-inositol treatment for ovulation induction, probably due to the presence of malabsorption caused by gut dysbiosis. The most recent evidence proposes dysbiosis and related chronic low-grade inflammation as the new DOGMA behind PCOS pathogenesis. In this regard, the recent findings on alpha-lactalbumin reports its effect in improving the absorption of different nutrients including myo-inositol as well as a crucial factor for reducing inflammation. Furthermore, this whey protein is well known for its effect as trophic agent for gastrointestinal flora in infants. For all these reasons, the investigators expect that the treatment with Inofolic HP (Myo-inositol and alpha-lactalbumin) will get an efficacy 20-25% higher than the treatment with inofolic.

ELIGIBILITY:
Inclusion Criteria:

* POCS women diagnosed using the Rotterdam Criteria

Exclusion Criteria:

* Amenorrhea (3 months)
* Other conditions causing ovulatory disorders and/or androgens hyper production such as: hyperprolactinemia, hypothyroidism, adrenal hyperplasia and Cushing syndrome
* Hormonal and/or pharmacological treatments in the previous 3 months that could interfere with ovulation
* Drastic changes in diet
* Treatment with product containing Myo-inositol in the previous 3 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
ovulation induction | after three months of treatment
  Ovulation indaction will by evaluated through ultrasound sonography

CONTACTS AND LOCATIONS:
Locations (1):
- Aleksandrovska University Hospital, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided